CLINICAL TRIAL: NCT05681156
Title: Curian S. Pneumo/Legionella Assay Beta Clinical Trial Protocol
Status: Completed | Type: Observational
Sponsor: Meridian Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN0015
Record Dates: First submitted 2022-12-27; First posted 2023-01-12 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Streptococcus Pneumoniae Infection; Legionella Pneumophila Serogroup 1 Infection
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients with suspected pneumonia: Leftover de-identified samples from standard of care will be taken from patients suspected of having pneumonia due to Streptococcus pneumoniae and/or Legionella pneumophila serogroup 1 infection.
  Interventions: Other: N/A- There is no intervention.

INTERVENTIONS:
Other: N/A- There is no intervention. — There is no intervention.

SUMMARY:
Beta trial to evaluate the preliminary clinical performance of the Curian S. pneumo/Legionella assay for its use in the qualitative detection of Streptococcus pneumoniae and/or Legionella pneumophila serogroup 1 antigens in human urine specimens.

DETAILED DESCRIPTION:
This study will evaluate the preliminary clinical performance of the RUO Curian S. pneumo/Legionella assay against two FDA cleared comparators for its use in the qualitative detection of Streptococcus pneumoniae and/or Legionella pneumophila serogroup 1 antigens in human urine specimens.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females, with symptom of pneumonia and for whom a Streptococcus pneumoniae and/or Legionella pneumophila serogroup 1 diagnostic test has been ordered by a practicing physician.
* At least 2mL of urine from fresh de-identified clinical specimen from standard of care lab testing
* Only one (1) specimen per patient will be included in the study
* Materials used within their expiration date
* Storage time and conditions within requested indications listed on RUO Package Insert

Exclusion Criteria:

* Specimens from patients for whom a Streptococcus pneumoniae and/or Legionella pneumophila serogroup 1 diagnostic test has not been ordered
* Storage times and conditions that exceed these study protocol requirements listed on RUO Package Insert
* Urine samples provided in unsatisfactory conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients arriving at hospital with suspected pneumonia
Sampling Method: Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
Agreement between Curian S. pneumo/Legionella Assay and two cleared FDA assays | 7 months
  Curian S. pneumo/Legionella Assay will be compared to the comparator assays (both FDA cleared)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided
No plan yet

REFERENCES:
- [Background] Yasuo S, Murata M, Nakagawa N, Kawasaki T, Yoshida T, Ando K, Okamori S, Okada Y; Japanese ARDS clinical practice guideline systematic review task force. Diagnostic accuracy of urinary antigen tests for pneumococcal pneumonia among patients with acute respiratory failure suspected pneumonia: a systematic review and meta-analysis. BMJ Open. 2022 Aug 11;12(8):e057216. doi: 10.1136/bmjopen-2021-057216. PMID 35953247
- [Background] Schimmel JJ, Haessler S, Imrey P, Lindenauer PK, Richter SS, Yu PC, Rothberg MB. Pneumococcal Urinary Antigen Testing in United States Hospitals: A Missed Opportunity for Antimicrobial Stewardship. Clin Infect Dis. 2020 Sep 12;71(6):1427-1434. doi: 10.1093/cid/ciz983. PMID 31587039